CLINICAL TRIAL: NCT06574932
Title: Screen Time and Sanity: The Impact of Multi-Strategy Approaches on Limiting Digital Exposure to Enhance Adolescent Mental Health
Brief Title: The Effect of Multi-Strategy Approaches on Limiting Digital Exposure
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Putra Malaysia (Other)
Collaborators: Green International University (Other)
Responsible Party: Principal Investigator, Arshed Muhammad, PhD studentship, Universiti Putra Malaysia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: FAHSS
Record Dates: First submitted 2024-08-25; First posted 2024-08-28 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Mental Health Wellness 1

STUDY DESIGN:
Intervention Model Description: Two-arm parallel design randomized control trial
Who Masked: Participant, Investigator
Masking Description: Participants and investigators will be blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The experimental group will be engaged in multi-strategy approaches including screen time and sanity challenges, weekly screen-free days, screen time reduction goals, screen time tracking, structured daily routines, parental involvement, and monitoring, family media plans, alternative engagements, and promotion of offline social interactions.
  Interventions: Behavioral: Multi-Strategic Approach
- Control (No Intervention): The control group will be given no intervention.

INTERVENTIONS:
Behavioral: Multi-Strategic Approach — The experimental group will be engaged in multi-strategy approaches including screen time and sanity challenges, weekly screen-free days, screen time reduction goals, screen time tracking, structured daily routines, parental involvement, and monitoring, family media plans, alternative engagements, and promotion of offline social interactions.
  Arms: Intervention group

SUMMARY:
In the digital age, university students are increasingly immersed in a technology-driven environment where smartphones, social media, and various digital platforms play a central role in their daily lives. While these technologies offer significant benefits, such as enhanced connectivity, access to information, and educational resources, they also pose potential risks to mental health. Excessive screen time, constant connectivity, and the pressure to maintain an online presence can lead to negative outcomes, including anxiety, depression, sleep disturbances, and reduced academic performance.

DETAILED DESCRIPTION:
Recent research highlights the growing concern over the impact of digital overuse on students' mental well-being. The constant barrage of notifications, the pressure to stay connected, and the addictive nature of social media can create a state of perpetual stress and distraction. This, in turn, can hinder students' ability to focus, engage in meaningful social interactions, and maintain a healthy balance between their academic and personal lives.

A multi-assignment program offers a promising intervention to counteract these negative effects. By encouraging students to disconnect from digital devices and reduce their online engagement temporarily, a digital detox can provide the opportunity to reset their relationship with technology. This period of disconnection allows students to regain control over their time, reduce stress, and foster healthier habits that support their mental well-being.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be enrolled as students at any of the three universities of Lahore.
* Participants should be 18 to 25 years old, as this demographic is typically more engaged in smartphone usage and may experience varying mental health effects.
* Participants must own and regularly use a smartphone. Regular use is a smartphone for at least two hours per day.
* Participants must be willing to provide written informed consent, acknowledging their understanding of the study and agreeing to participate voluntarily.
* Participants must be able to read and understand the language in which the questionnaires and assessments are administered (likely English or Urdu, depending on the study design).
* Only full-time students will be included to ensure that their daily routines and stress levels are more comparable across the study group.

Exclusion Criteria:

* Individuals who have been diagnosed with severe psychiatric disorders (such as schizophrenia, bipolar disorder, or other major psychiatric conditions) will be excluded. These conditions could introduce confounding variables that may affect the study's results.
* Individuals who are currently undergoing treatment for severe mental health conditions or are taking medication that could significantly impact mental health and smartphone usage will be excluded to avoid confounding effects.
* Individuals who have recently experienced major life events (such as the death of a close family member, major accidents, or other significant trauma) within the last six months may be excluded, as these events could influence mental health independently of smartphone use.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 700 (Estimated)
Dates: Start 2024-08-27 (Estimated); Primary Completion 2025-04-15 (Estimated); Study Completion 2025-05-10 (Estimated)

PRIMARY OUTCOMES:
Generalized anxiety | 6-months from baseline
  Generalized anxiety change will be measured by (GAD-7). seven-item instrument that is used to measure or assess the severity of generalized anxiety disorder (GAD). The GAD-7 score is calculated by assigning scores of 0, 1, 2, and 3, to the response categories of "not at all," "several days," "more than half the days," and "nearly every day," respectively, and then adding together the scores for the seven questions. GAD-7 total score for the seven items ranges from 0 to 21.Score 0-4: Minimal Anxiety. Score 5-9: Mild Anxiety. Score 10-14: Moderate Anxiety. Score greater than 15: Severe Anxiety.

SECONDARY OUTCOMES:
Depression | 6-months from baseline
  Depression change will be measured by PHQ-9. PHQ-9 scores can be used to plan and monitor treatment. To score the instrument, tally the numbers of all the checked responses under each heading (not at all=0, several days=1, more than half the days=2, and nearly every day=3). Add the numbers together to total the score on the bottom of the questionnaire. PHQ-9 comprises five categories, where a cut-off point of 0-4 indicates no depressive symptoms, 5-9 mild depressive symptoms, 10-14 moderate depressive symptoms, 15-19 moderately-severe depressive symptoms, and 20-27 severe depressive symptoms

CONTACTS AND LOCATIONS:
Overall Officials: MUHAMMAD ARSHED, PhD, Principal Investigator — University of Lahore

IPD SHARING:
Plan to Share IPD: No
The study protocol, statistical plan, and results will be disseminated through publications in peer-reviewed Journals.

REFERENCES:
- [Background] Shakya HB, Christakis NA. Association of Facebook Use With Compromised Well-Being: A Longitudinal Study. Am J Epidemiol. 2017 Feb 1;185(3):203-211. doi: 10.1093/aje/kww189. PMID 28093386
- [Background] Basen I. You can't stop checking your phone because Silicon Valley designed it that way. CBC Radio 2018 Sept 14. Available: www.cbc.ca/radio/thesundayedition/the-sunday-edition-september-16-2018-1.4822353/you-can-t-stop-checking-your-phone-because-silicon-valley-designed-it-that-way-1.4822360
- [Background] NHS Digital. Mental Health of Children and Young People in England, 2017: Summary of key findings. NHS Digital; 2018 [cited 2019 Sep 21]. Available from: https://files.digital.nhs.uk/A6/EA7D58/MHCYP%202017%20Summary.pdf
- [Background] Patalay P, Gage SH. Changes in millennial adolescent mental health and health-related behaviours over 10 years: a population cohort comparison study. Int J Epidemiol. 2019 Oct 1;48(5):1650-1664. doi: 10.1093/ije/dyz006. PMID 30815691
- [Background] Mojtabai R, Olfson M, Han B. National Trends in the Prevalence and Treatment of Depression in Adolescents and Young Adults. Pediatrics. 2016 Dec;138(6):e20161878. doi: 10.1542/peds.2016-1878. Epub 2016 Nov 14. PMID 27940701